CLINICAL TRIAL: NCT06534554
Title: Improving Gout Care After an Emergency Department Visit for Acute Gout
Brief Title: Improving Gout Care After an ED Visit
Acronym: CARE-Gout
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Kenneth Saag, MD, MSc, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 300004983-053; 000541304 (Other Grant/Funding Number: Horizon Therapeutics)
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Patient Navigation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Navigation (Experimental): A lay patient navigator will contact patients seen in the UAB ED via phone within ~72 hours following the ED visit. During this initial phone conversation, the navigators will: 1) conduct a baseline assessment to identify barriers to attending an outpatient visit for gout care and to adhering to gout treatment recommendations and 2) determine the level of support and assistance needed by the patient.
  Interventions: Behavioral: Patient Navigation
- Control (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Patient Navigation — A lay patient navigator working will contact patients seen in the UAB ED via phone within ~72 hours following the ED visit. During this initial phone conversation, the navigators will: 1) conduct a baseline assessment to identify barriers to attending an outpatient visit for gout care and to adhering to gout treatment recommendations and 2) determine the level of support and assistance needed by the patient.
  Arms: Patient Navigation

SUMMARY:
The prevalence of gout has been steadily increasing over several decades and is correlated with the rising burden of obesity, chronic cardiac and renal disease; all conditions overrepresented in the Southeastern U.S. - particularly in African Americans. Through a novel post-emergency department visit intervention, we aim to improve the care patients with gout receive, both during acute exacerbations and long-term. A secondary goal of the project is to concurrently enhance participation of minorities in biomedical research in the Deep South.

DETAILED DESCRIPTION:
The prevalence of gout has been steadily increasing and is correlated with the rising burden of obesity, chronic cardiac and renal disease; all conditions overrepresented in the Southeast U.S. - particularly in African Americans. Many patients with acute gout receive care at the emergency department (ED), particularly underserved urban populations in the Deep South. Appropriate outpatient follow-up for an acute flare after an ED visit is variable. Indeed, in a preliminary analysis of a retrospective cohort study of patients with acute gout treated at our urban medical center ED, only 46% of patients followed up with an outpatient clinician in our healthcare system within 6 months of their ED visit. Even fewer (36%) had an outpatient visit specifically addressing gout care within 6 months post-ED visit. This population of patients that seek acute gout care in the ED represent an important group that may benefit from interventions focused on improving gout quality of care, such as promoting outpatient follow-up.

While having a mechanism to identity acute gout patients in the ED is fundamental for enhancing care for patients with acute gout, recruiting people with acute gout who receive care in the ED outside regular business hours is challenging. One potential solution involves approaching patients after their ED visits remotely using patient navigators. The 36-72 hour period after their ED visit represents a critical time during which patients may be more receptive to efforts focused on improving healthy behaviors including scheduling outpatient follow-up (i.e., a "teachable moment). Patient navigators are trained, lay individuals of similar cultural background, and region, who provide personal guidance to patients and engage "hard-to-reach" groups, reduce access barriers, and encourage healthy behaviors such as engaging in outpatient chronic disease management.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Able to communicate and understand English or Spanish
* Confirmed acute gout flare by EMR review at ED visit

Exclusion Criteria:

* Enrollment in an ongoing RCT (NCT04075903) testing a behavioral intervention employing "storytelling".

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Follow-Up Visit Addressing Gout within 3 Months | 3 months
  Proportion of patients that have a follow-up visit addressing gout in the 3-month period after the ED visit.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No